CLINICAL TRIAL: NCT06529640
Title: Can a Periosteal Pedicle Flap Replace the Subepithelial Connective Tissue Graft in the Management of Gingival Recession? Randomized Controlled Clinical Trial
Brief Title: Periosteal Pedicle Flap Versus Subepithelial Connective Tissue Graft in Management of Gingival Recession
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Alzahraa Alghriany, Lecturer, Oral medicine, Periodontology and Oral diagnosis, Faculty of dentistry, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: periosteal pedicle flap
Record Dates: First submitted 2024-07-26; First posted 2024-07-31 (Actual); Last update posted 2024-07-31 (Actual); Status verified 2024-07

CONDITIONS: Gingival Recession
MeSH Terms: conditions — Gingival Recession

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Subepothelial connective tissue graft (SCTG) group (Active Comparator): Subepithelial connective tissue graft from palate then coronally positioning flap to cover root recession
  Interventions: Procedure: SCTG followed by coronally postionting flap
- Periosteal pedicle flap (PPF) group (Active Comparator): periosteal flap elevation and repositioning to the root then coronally positioning flap to cover root recession
  Interventions: Procedure: periosteal flap followed by coronally postionting flap

INTERVENTIONS:
Procedure: SCTG followed by coronally postionting flap — The SCTG will be harvested from the palate followed by coronally postionting flap
  Arms: Subepothelial connective tissue graft (SCTG) group
Procedure: periosteal flap followed by coronally postionting flap — he periosteal pedicle graft obtained is then turned over the exposed root surface then followed by coronally postionting flap
  Arms: Periosteal pedicle flap (PPF) group

SUMMARY:
Gingival recession is defined as the apical shift of the marginal gingiva from its normal position on the crown of the tooth to levels on the root surface beyond the cemento-enamel junction (CEJ).Various surgical procedures including repositioned flaps as well as autogenous and other type grafts have been used in the treatment of gingival recession.The present gold standard technique is the bilaminar technique using the subepithelial connective tissue graft (SCTG) which provides for long-term stability but also increases tissue morbidity.Hence, a suitable alternative technique - the periosteal pedicle flap (PPF) - has been practiced, which is less invasive, does not require a second surgical site, and provides a graft of adequate dimensions.

ELIGIBILITY:
Inclusion Criteria:

* Patients with one or more Miller's Class 1 and Class II buccal recessions demonstrating ≤20% of plaque and bleeding scores, respectively, after Phase I therapy.
* age from 18 th 60 years.

Exclusion Criteria:

* Smokers
* patients with malposed or crowded teeth
* pregnant and lactating women
* patients using medications that could affect the periodontal status

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 10 (Estimated)
Dates: Start 2024-08-01 (Estimated); Primary Completion 2024-11-01 (Estimated); Study Completion 2024-11-01 (Estimated)

PRIMARY OUTCOMES:
the percentage of root coverage (%RC) | at base line, 1 month and 3 months after treatment
  to measure the coverage percentage of root recession by UNC periodontal probe Preoperative recession depth - Postoperative recession depth /Preoperative recession depth x 100

SECONDARY OUTCOMES:
recession depth | at base line, 1 month and 3 months after treatment
  to measure vertical recession by UNC periodontal probe from cemento-enamel junction (CEJ) to the gingival margin.
recession width | at base line, 1 month and 3 months after treatment
  to measure horizontal recession by UNC periodontal probe the distance between the CEJ and the gingival margin
clinical attachment gain | at base line, 1 month and 3 months after treatment
  to measure the periodontal attachment gain after treatment by UNC periodontal probe subtracting the sulcus depth from the distance between the free gingival margin and the mucogingival junction.
keratinized tissue gain | at base line, 1 month and 3 months after treatment
  measure the gain in keratinized gingivaby UNC periodontal probe from the most apical point of the gingival margin to the mucogingival junction (MGJ) at the middle buccal point.